CLINICAL TRIAL: NCT05722808
Title: What is the Rate of Surgical Treatment in Adult Patients With Displaced Distal Radius Fractures Managed According to the Danish National Clinical Practice Guidelines? - A Single Center Retrospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2214020
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Distal Radius Fracture
Keywords: Distal radius fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Through this study we aim to investigate the rate of DRFs initially treated with successful closed reduction (to an acceptable position, then immobilized in a plaster cast), that re-displace and end up requiring surgery.

This study will clarify the incidence of DRFs where surgical intervention could potentially be avoided if the initial closed reduction lasted until sufficient bone healing was attained. As DRFs are the most common fracture of the adult population treated in the Danish emergency departments, the aim of this study is to examine the amount of people with DRFs that could potentially avoid surgery and thereby lowering the cost to the health care system, as well as save the patient invasive surgery. Furthermore, we expect to classify which specific types of fractures according to Arbeitsgemeinschaft für Osteosynthesefragen/ Orthopaedic Trauma Association (AO/OTA) classification system have a high or low incidence of secondary surgery after primary closed reduction.

DETAILED DESCRIPTION:
Study rational Only a limited number of orthopedic national clinical practice guidelines (NCPG) exist in Denmark. In 2013 a NCPG regarding the treatment of distal radius fractures (DRFs) was introduced in Denmark [1]. Without any major changes, it was updated in 2017, which is the latest version. Displaced distal radius fractures are very frequent in the adult population, with about 20.000 fractures pr. year, and the incidence is still increasing as the population ages [1, 2]. Two-thirds of DRFs in adults are displaced and require closed reduction [5]. Unfortunately, a large number of the reduced DRFs (32-64%) re-displace during cast immobilization within the first weeks after reduction [1]. According to the NCPG, it is considered good clinical practice to offer surgical treatment to patients of any age if a conventional wrist X-ray examination, following reduction of the fracture, reveals one or more of the radiological parameters described in figure 1. Furthermore, it is described as good clinical practice to be cautious about offering surgery to any patient with a low functional level, regardless of their age [1].

Background Each year about 20.000 adult patients are treated for DRF in the Danish emergency departments across the country [1]. Therefore, the DRF is the most frequently treated fracture among adults in the Danish healthcare system. As the population ages the number of DRF increases. Furthermore, the rate of surgical treatment of DRF increases independently, probably due to an international change towards more interventional treatment, favoring surgery above conservative treatment.

The years up to 2013, a change was observed in the surgical method concerning treatment of DRF. Internal fixation with a volar plate and screws increased at the expense of K-wires or external fixation. This change is seen even based on sparse literature evidence [1].

In the general population, the distribution of DRFs is bimodal, with the incidence peaks in young men - due to high energy trauma - and in postmenopausal women [2]. The majority of DRFs in the second group are caused by a fall on an outstretched hand from one's upright position, thus it is considered low-energy fractures. There is a significant predominance of women to whom this type of fracture occurs, which is connected to the fact that osteoporosis is an underlying cause [1]. In a Swedish study, Rundgren et al. found that 78% of all DRFs occurred in women [2], while it was found in a British study that the rate of women to men was 68:38 [3].

What does this trial add to current knowledge? Through this study we aim to investigate the rate of DRFs initially treated with successful closed reduction (to an acceptable position, then immobilized in a plaster cast), that re-displace and end up requiring surgery.

This study will clarify the incidence of DRFs where surgical intervention could potentially be avoided if the initial closed reduction lasted until sufficient bone healing was attained. As DRFs are the most common fracture of the adult population treated in the Danish emergency departments, the aim of this study is to examine the amount of people with DRFs that could potentially avoid surgery and thereby lowering the cost to the health care system, as well as save the patient invasive surgery. Furthermore, we expect to classify which specific types of fractures according to Arbeitsgemeinschaft für Osteosynthesefragen/ Orthopaedic Trauma Association (AO/OTA) classification system have a high or low incidence of secondary surgery after primary closed reduction.

Hypothesis We estimate the rate of surgical intervention of DRFs initially reduced to an acceptable position to be above 40%.

Aim The primary objective is to assess the rate of surgical treatment in adult patients with distal radial fractures, initially reduced successfully, managed in a single center according to the danish national clinical practice guidelines (NCPG).

Primary endpoint The purpose of this study, is to determine the frequency of secondary displacement of DRFs, initially treated with closed reduction and casting, but subsequently resulting in secondary surgery.

Secondary endpoints

* We aim to compare the rate of DRF displacement following primary closed reduction found in this study with a similar cohort treated in the Netherlands [4].
* We will perform a sub analysis of risk of secondary displacement according to the "Arbeitsgemeinschaft für Osteosynthesefragen" (AO) classification system for DRFs.
* We will determine the frequency of DRFs with unacceptable position, according to NCPG, following initial reduction that are treated non-surgical.
* We will determine the number of reductions performed at the initial visit in the emergency department following a distal radius fracture per patient.

Study Design This study will be conducted as a retrospective cohort study. In addition, outcomes from this study will be compared to outcomes from a comparable cohort from a previous retrospective study conducted in the Netherlands.

Population Adult patients with displaced DRFs treated at North Zealand Hospital (Nordsjællands Hospital, NOH) from 1.1.2018 to 31.12.2019.

Inclusion criteria Adult patients (≥18 years) with a DRF (DS252, DS252A, DS252B, DS252C and DS526), treated in the emergency department at NOH.

Exclusion criteria

* Concomitant fracture of the ulna (except ulnar styloid process' fractures)
* Non-displaced DRFs
* Multiple trauma patients
* Ipsilateral upper extremity fractures, interfering with the treatment of the DRF Method Data will be retrieved from the electronic patient records (Sundhedsplatformen (SP)). Potential participants will be identified by relevant diagnosis codes (DS252, DS252A, DS252B, DS252C and DS526), treated in the emergency department at NOH with closed reduction and an immobilizing cast from Jan 1st 2018 to Dec 31st 2019. We expect to include approximately 750 participants.

Data relevant to the above-described outcomes (i.e radiologic data, diagnosis/procedure codes and information from outpatient clinic visits) and data relevant for baseline characteristics will be extracted from patient electronic journals and transferred to investigators.

All extracted data will be transferred in pseudonymized form to an on-line data capturing system (REDCAP).

A team of orthopedic surgeons from the orthopedic department, NOH, will be asked to assess radiographic images from the initial visit to the emergency department to assess:

* Classification according to AO
* Non-displaced yes/no
* Radiographic measurements according to https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4641087/ (radial shortening, ulnar variance and volar/dorsal angulation)

A comparable cohort from an ongoing prospective study of DRFs, performed in the Netherlands, has been identified and the responsible researcher has been contacted and agreed to provide data for a comparison of data between the two groups. Data will be transferred in anonymized form to the primary investigator of this study and stored at a secure drive. The primary and secondary outcomes outlined above will be compared across the two cohorts.

Due to the study design, it will be possible to repeat the study in other hospitals and compare the results across the Danish emergency departments as well as international.

Statistical analysis Rate of DRF displacement, following initial reduction and cast treatment, is described with summary statistics.

Categorical and ordinal variables will be presented in percentages of the analyzed group. Continuous variables will be presented as mean followed by standard deviation. If continuous variables were not normally distributed, they will be presented as median with (25% and 75% quartiles) and log transformed before further analysis.

Categorical and ordinal variables are compared across groups using χ2 test (Pearson test). If a low number of expected frequencies is encountered, Fisher's exact test is used. For analysis of differences in continuous variables between groups, t-test will be carried out.

Multiple regression will be performed to identify possible associations between relevant clinical variants and risk of DRF displacement following initial reduction and cast treatment.

All statistical analyses will be performed in the SAS ® Studio 3.7 (SAS Institute Inc., Cary, NC, USA).

Statistical significance is defined as a probability (p-value) lower than 5%. Perspective The results of this study will allow us to clarify the number of patients with DRF where surgery could potentially be avoided. If a specific group of patients (determined radiologically due to AO-classifications) with larger risk of DRF displacement following initial reduction and cast treatment is identified, there would be a great incentive to improve the treatment of this group. In addition, the comparison with a cohorte from the Netherlands will allow us to identify international differences in treatment and diagnosis of DRFs. The results of this study may eventually lead to a reduction in surgical treatment of DRFs and thereby a possible reduction in cost in relation to DRF treatment to the society.

Quality control and monitoring The study will be conducted in accordance with the Helsinki declaration on "Ethical Principles for Medical Research Involving Human Subjects". The principles of Good Clinical Practice were followed throughout the study.

The STROBE guidelines will be followed in the initiation, data handling and presentation of the study.

The study protocol will be registered in the "The ISRCTN registry" before initiation.

No monitoring of the study is needed or planned of this retrospective cohort study. As the radiographic data for each patient has been evaluated by orthopedic consultant or senior registrar at least three times (initially in emergency department, day after at conference, in out-patient clinic and/or in the operating theater), we deem it highly unlikely that any new findings of clinical relevance should happen. In the unlikely event that a new clinical finding should be done we will consult the local radiograph responsible for orthopedic radiology at NOH.

Ethical considerations and data safety To protect the patient's privacy and integrity, data will be extrapolated from SP and pseudonymized, and it will not be possible to identify the individuals. This study will not have any effect on the treatment or outcome for the patient cohort, but will solely help to identify improvements of future treatments. This study will investigate potential areas of DRF treatment where improvement can be made to potentially avoid surgery in this large fragile population.

Ethical committee approval Before the study is initiated, approval from relevant ethical and data security agencies will be attained; "National Videnskabsetisk Komite, "Sundhedsdatastyrelsen, Forskerservice" and the Danish Data Protection Agency https://sundhedsdatastyrelsen.dk/da/forskerservice/ansog-om-data.

Recruitment As this is a retrospective cohort study there is no need to recruit patients, as the data needed can be found in the electronic patient records.

Economy There is no funding for this project, as well as no sponsors or donors. The primary investigator and all secondary investigators are unpaid and perform the investigation in their spare-time. Except the clinically responsible investigator, Jonas Askø Andersen, who is head of research in the Orthopedic department in North Zealand Hospital.

Dissemination of results We expect to complete the data- and statistical analysis in September 2022. At this point the data and conclusion will be published in an international or national peer-reviewed medical journal. Both positive, negative and inconclusive data will be published. In addition, data from the study will be presented at national and international conferences if possible. Should publication in a peer-reviewed journal not be possible, data will be published in an open access database.

Patient information As this study does not add new treatments or diagnostic methods to the patients involved and does not use individual or patient identifiable data, we have applied for data access without written consent from included individuals and therefore patient information has been deemed unnecessary.

References

1. https://www.sst.dk/-/media/Udgivelser/2014/NKR-H%C3%A5ndledsn%C3%A6re-underarmsbrud/National-clinical-guideline-on-the-treatment-of-distal-radial-fractures.ashx?sc_lang=da&hash=A867AD76B6ECFF5A7307A0C006E0938A
2. Rundgren J, Bojan A, Navarro CM et. al., "Epidemiology, classification, treatment and mortality of distal radius fractures in adults: an observational study of 23,394 fractures from the national Swedish fracture register", BMC Musculoskeletal Disorders (2020) 21:88,
3. Stirling ERB, Johnson NA, Dias JJ. Epidemiology of distal radius fractures in a geographically defined adult population. J Hand Surg Eur Vol. 2018;43(9):974-82.
4. Berger AC , Barvelink B, Reijman M et. al., "Does circumferential casting prevent fracture redisplacement in reduced distal radius fractures? A retrospective multicentre study", Journal of Orthopaedic Surgery and Research (2021) 16:722
5. Brogren E, Petanek M and Atroshi I, "Incidence and characteristics of distal radius fractures in a southern Swedish region", BMC Musculoskeletal Disorders

ELIGIBILITY:
Inclusion criteria Adult patients (≥18 years) with a DRF (DS252, DS252A, DS252B, DS252C and DS526), treated in the emergency department at North Zealand Hospital.

Exclusion criteria

* Concomitant fracture of the ulna (except ulnar styloid process' fractures)
* Non-displaced DRFs
* Multiple trauma patients
* Ipsilateral upper extremity fractures, interfering with the treatment of the DRF

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with displaced DRFs treated at North Zealand Hospital from 1.1.2018 to 31.12.2019.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of surgical treatment | Anticipated to be completed by 31/05-2023
  Rate of surgical treatment of distal radial fractures treated at North Zealand Hospital

SECONDARY OUTCOMES:
Rate of fracture displacement following primary conservative treatment compared with Dutch cohort | Anticipated to be completed by 31/05-2023
  Comparison of the rate of DRF displacement following primary closed reduction found in this study with a similar cohort treated in the Netherlands
sub analysis of risk of secondary displacement according to the "Arbeitsgemeinschaft für Osteosynthesefragen" (AO) classification system for DRFs | Anticipated to be completed by 31/05-2023
Incidence of distal radial fractures with unaccetable displacement following following initial reduction | Anticipated to be completed by 31/05-2023
  Analysis of the frequency of distal radial fractures with unacceptable position, according to danish national guidelines, following initial reduction that are treated non-surgical
Number of reductions performed per patient with distal radial fractures | Anticipated to be completed by 31/05-2023

CONTACTS AND LOCATIONS:
Locations (1):
- North Zealand Hospital, Hillerød, Denmark